CLINICAL TRIAL: NCT02140372
Title: Anti-platelet Effects of Colchicine in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S13-00747
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: colchicine; platelet activity; neutrophil
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Volunteer group (Experimental): Baseline blood draw followed by colchicine followed by blood draw 2 hours and 24 hours later
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — Colchicine 1.2 mg followed by 0.6 mg one hour later
  Other Names: Colcrys

SUMMARY:
This is a pilot study. Volunteers will be given 1.8 mg (1.2 mg followed by 0.6 mg one hour later), 1.2 mg, or 0.6 mg of colchicine. Blood will be collected prior to drug administration, 2 hours after colchicine administration, and 24 hours after colchicine administration via the antecubital vein and evaluated for markers of platelet activity and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be more than 18 years of age

Exclusion Criteria:

1) history of cardiovascular disease, including myocardial infarction, history of percutaneous coronary angioplasty or stent, peripheral vascular disease or stroke; 2) history of myelodysplasia; 3) medications known to affect platelet function, including non-steroidal anti-inflammatory drugs, antihistamines, and selective serotonin reuptake inhibitors, during the 5 days prior to participation; 4) medications known to interact with colchicine; 5) history of intolerance to colchicine; 6) acute or chronic symptoms of diarrhea, nausea, or vomiting within 1 month prior to enrollment; 7) known anemia or hemoglobin <10mg/dL; 8) platelet count <100,000 or > 450,000; 9) creatinine clearance <30cc/minute; 10) any known hemorrhagic diathesis; 11) pregnant; 12) Unable to consent; or 13) Participating in a competing study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, MS, Principal Investigator — NYU SOM
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Volunteer Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Volunteer Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Monocyte Platelet Aggregate: Baseline
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: percentage of monocyte-platelet aggregat
Arm/Group | Volunteer Group
Number analyzed (Participants) | 10
percentage of monocyte-platelet aggregat | 27.8 [21.6 to 57.3]

2. Secondary Outcome: Light Transmission Aggregometry: Baseline
Description: In response to adenosine diphosphate
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: percentage of max platelet aggregation
Arm/Group | Volunteer Group
Number analyzed (Participants) | 10
percentage of max platelet aggregation | 48.7 [33.5 to 85.3]

3. Primary Outcome: Monocyte Platelet Aggregate: 2 Hours
Time Frame: 2 Hours
Measure: Median (Inter-Quartile Range); unit: percentage of monocyte-platelet aggregat
Arm/Group | Volunteer Group
Number analyzed (Participants) | 10
percentage of monocyte-platelet aggregat | 22 [19.0 to 30.8]

4. Secondary Outcome: Light Transmission Aggregometry: 2 Hours
Description: In response to adenosine diphosphate
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: percentage of max platelet aggregation
Arm/Group | Volunteer Group
Number analyzed (Participants) | 10
percentage of max platelet aggregation | 66.6 [23.6 to 87.3]

5. Secondary Outcome: Light Transmission Aggregometry: Baseline
Description: In response to adenosine epinephrine
Time Frame: baseline
Measure: Median (Inter-Quartile Range); unit: percentage of max platelet aggregation
Arm/Group | Volunteer Group
Number analyzed (Participants) | 10
percentage of max platelet aggregation | 84.9 [61.8 to 90.2]

6. Secondary Outcome: Light Transmission Aggregometry: 2 Hours
Description: In response to adenosine epinephrine
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: percentage of max platelet aggregation
Arm/Group | Volunteer Group
Number analyzed (Participants) | 10
percentage of max platelet aggregation | 84.6 [48.6 to 87.7]

7. Secondary Outcome: Platelet Adhesion: Baseline
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: percentage of adhered platelets
Arm/Group | Volunteer Group
Number analyzed (Participants) | 10
percentage of adhered platelets | 10.2 [2.5 to 32.6]

8. Secondary Outcome: Platelet Adhesion: 2 Hours
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: percentage of adhered platelets
Arm/Group | Volunteer Group
Number analyzed (Participants) | 10
percentage of adhered platelets | 2.0 [0.2 to 9.5]

ADVERSE EVENTS:
Arm/Group | Volunteer Group
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes